CLINICAL TRIAL: NCT05491629
Title: Perceptıons Of The Surgıcal Team Regardıng The Competencıes Of The Operatıng Room Nurse And Factors Affectıng The Competence
Brief Title: Competencies of Operating Room Nurses and Influencing Factors
Status: Completed | Type: Observational
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Öğr. Gör. Ayşe UÇAK, Principal Investigator, Burdur Mehmet Akif Ersoy University
Other Study IDs: AUCAK
Record Dates: First submitted 2022-07-07; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Competence; Nurse's Role
Keywords: Operating room nursing, competence, competency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgical team members: The aim of this study is to determine with a deep understanding the perceptions of the operating room nurses' competence and the surgical team's views on the competence of nurses and the factors affecting them. In the research, parallel data type in convergent parallel mixed design (convergent parallel) was used to obtain rigorous, valid and reliable data with survey questions and individual interviews. In the quantitative dimension of the study, it was aimed to determine the perceptions of the operating room nurses about their competencies, and in the qualitative aspect, the thoughts/opinions of the entire surgical team about the competency of the operating room nurses and the factors affecting them.
  Interventions: Other: type of parallel data in a convergent parallel hash pattern (near time)

INTERVENTIONS:
Other: type of parallel data in a convergent parallel hash pattern (near time) — The quantitative part of the study is a descriptive study with the Perceived Perioperative Competence Scale-Revised to determine the perceptions of operating room nurses about their competencies.
  It is a case study in order to reveal the opinions of the surgical team members about the competencies of the operating room nurses and the affecting factors through individual in-depth interviews and to better explain the current situation at the qualitative stage, which is carried out simultaneously.

SUMMARY:
Aim: The aim of this study was to determine the perceived competence of operating room nurses and the opinions of the surgical team, regarding the competence of nurses and the influencing factors with a deep understanding.

Method: This convergent parallel mixed-methods study was carried out with members of the surgical team working in 17 hospitals including three public, two university, one city, one education and research, and ten private ones located in city center of Burdur, Isparta and Antalya provinces. The data were collected between May 1th, 2020 and August 20th, 2020 using Quantitative and Qualitative Personal Information Forms, Perceived Perioperative Competence Scale (PPCS-R) and semi-structured interview form. The quantitative data were assessed using the SPSS 24.0 package program, and the qualitative data were assessed using content analysis and thematic analysis. The quantitative and qualitative data were analyzed independently, and interpreted based on analytical generalization in the discussion section.

DETAILED DESCRIPTION:
Aim: The aim of this study was to determine the perceived competence of operating room nurses and the opinions of the surgical team, regarding the competence of nurses and the influencing factors with a deep understanding.

Method: This convergent parallel mixed-methods study was carried out with members of the surgical team working in 17 hospitals including three public, two university, one city, one education and research, and ten private ones located in city center of Burdur, Isparta and Antalya provinces. The sample of the quantitative dimension of the study consisted of 224 operating room nurses working in authorized institutions, and the qualitative dimension consisted of 54 team members including 21 operating room nurses, 21 surgeons, 3 anesthesiologists, and 9 technicians/operators. The data were collected between May 1th, 2020 and August 20th, 2020 using Quantitative and Qualitative Personal Information Forms, Perceived Perioperative Competence Scale (PPCS-R) and semi-structured interview form. The quantitative data were assessed using the SPSS 24.0 package program, and the qualitative data were assessed using content analysis and thematic analysis. Quantitative data were analyzed using descriptive analysis, ANOVA, Mann Whitney U and Kruskal-Wallis H tests. Qualitative data were assessed through descriptive content analysis. The quantitative and qualitative data were analyzed independently, and interpreted based on analytical generalization in the discussion section.

ELIGIBILITY:
Inclusion Criteria:

* Quantitative At least six months of operating room experience nurses Qualitative At least six months of operating room experience surgical team members

Exclusion Criteria:

Willingness to withdraw from the study at any time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The universe of the research consists of the hospitals located in the city centers of Burdur, Isparta and Antalya in the Western Mediterranean Region. The sample consists of surgical team members working in the operating rooms of 17 hospitals, two of which are university, one is research practice, four are state and ten are private.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
competence Factors affecting the competence of operating room nurses | 6 week
  In the quantitative dimension of the study, the competency areas of operating room nurses were evaluated in 6 dimensions with the revised perioperative competency scale. The factors of the scale included "foundational knowledge and skills" (9 items), "leadership" (8 items), "collaboration" (6 items), "proficiency" (6 items), "empathy" (5 items), and "professional development" (6 items). In the qualitative aspect of the research, individual in-depth interviews with the surgical team members were made by descriptive and content analysis, and competency areas were determined.
  security non-technical arae

SECONDARY OUTCOMES:
factors | 6 week
  In the quantitative aspect of the study, the Perceived Perioperative Competence Scale-Revised and the sociodemographic characteristics of nurses were compared.
  In the qualitative aspect of the study, descriptive and content analysis were made in the interviews with the members of the surgical team and the influencing factors were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Uçak-lecturer, Principal Investigator — Akdeniz University
Locations (1):
- Fatma Cebeci, Muratpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided